CLINICAL TRIAL: NCT07054216
Title: Efficacy of a Probiotic on Gut Health, Immune Maturation, and Well-being in Term Newborns - a Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Probiotic for Infants
Acronym: BABIES II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Chr Hansen (Industry)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Professor Andreas Munk Petersen, MD, PhD, DMSc, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HND-IN-057; H-25028285 (Other: Ethics Committee Case number)
Record Dates: First submitted 2025-06-13; First posted 2025-07-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy Infants
Keywords: Infant; Gastrointestinal Microbiome; Diet, Food, and Nutrition
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial in term newborns with an 8½ months intervention period from 14 days of age until 9 months of age followed by a 3 months short-term follow-up period until 1 year of age and a long-term follow-up until 18 years of age
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic Dietary supplement
  Interventions: Other: Probiotic
- Placebo (Placebo Comparator): Identical looking placebo consisting of maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Other: Probiotic — Given daily from 14 days of age until 9 months of age
  Arms: Probiotic
Dietary Supplement: Placebo — Given daily from 14 days of age until 9 months of age
  Arms: Placebo

SUMMARY:
The BABIES II study is a single-center, randomized, double-blinded, placebo-controlled study in newborns with an 8½ months intervention period from 14 days of age to 9 months of age followed by a 3-months short-term follow-up period until 1 year of age and a possible long-term follow-up until 18 years of age. The study will evaluate the effect of supplementation with a probiotic strain on different health outcomes.

ELIGIBILITY:
"Inclusion Criteria"

Inclusion Criteria for the pregnant person

1. Pregnant person above 18 years of age in gestational week 36+0-38+0 (at Visit 0)
2. Singleton pregnancy
3. Ability to read and speak Danish
4. Plan to breastfeed
5. Provided voluntary written informed consent.

Inclusions Criteria for the newborn

1. Born at full-term ≥37+0
2. Birth weight ≥ 2500 g
3. APGAR score of ≥ 7 within the first 5 min of life.

"Exclusion Criteria" Exclusion Criteria for the pregnant person

1. Pregnancy at 38 weeks + 0 or later at the time of recruitment
2. Pregnancy with significant fetal abnormality at ultrasound scan of the fetus at gestational age 19-20 weeks
3. Alcohol or drug abuse
4. Plan to give birth at other hospitals than Copenhagen University Hospital Hvidovre
5. Pregnant person with any contraindications for breastfeeding.

Exclusion Criteria for the newborn

1. Congenital disorders that could affect their safety or the study outcome
2. Admission to Neonatal Intensive Care Unit for more than 24 hours
3. Participation in another clinical intervention study which can interfere with this probiotic intervention
4. Probiotics other than the study product.

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 378 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Total abundance of Bifidobacteria | At 3 months of age
  Abundance of Bifidobacteria in infant fecal samples by quantitative PCR

SECONDARY OUTCOMES:
Infant fecal pH | Birth (first stool after meconium), 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, and 1 year
  Changes in Fecal pH measured in fecal water from fecal samples
Infant gut microbiome composition | Birth (first stool after meconium), 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, and 1 year
  Changes in gut microbiome composition analyzed by metagenomics analysis of fecal stool samples (shotgun DNA sequencing)
Proportion of infants with hard or very hard stool consistency | 4 months, 5 months, 6 months
  The proportion of infants with episodes 'hard' and/or 'very hard' stool consistency assessed as the difference in numbers of infants who experience 'hard' and /or 'very hard' stool consistency during weaning (from first introduction of solid food) between the two groups

OTHER OUTCOMES:
Infant gut metabolome composition | Birth (first stool after meconium), 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, and 1 year
  Changes in the overall infant fecal metabolome assessed by untargeted metabolomics
Quantity of metabolites in infant fecal samples | Birth (first stool after meconium), 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, and 1 year
  Quantification of metabolites in infant fecal samples measured by targeted metabolomics
Infant Whole Gut Transit Time | 9 months and 1 year
  Whole gut transit time measured by sweet corn test
Abundance of clinically relevant pathogens in feces | Birth (first stool after meconium), 2 weeks, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, and 1 year
  Abundance of clinically relevant pathogens in feces (e.g., but not limited to Staphylococcus aureus, Staphylococcus epidermidis, Staphylococcus haemolyticus, Pseudomonas aeruginosa, Enterobacter, Klebsiella, Proteus, group B Streptococcus, Clostridioides difficile, Bacillus subtilis and Acinetobacter measured by DNA/RNA sequencing of fecal samples
Infant bowel habits | Weekly (0-52 weeks of age)
  Changes in bowel habits as measured by stool frequency and stool consistency. The consistency will be assessed by a modified Diapered Infant Stool Scale continuously in an electronic diary weekly from birth to 1 year of age
Pediatric Quality of Life Inventory™ 2.0 Family Impact Module (PedsQL™) | 3 months, 6 months, 9 months, and 1 year
  Familys health-related quality of life will be measured by Pediatric Quality of Life Inventory™ 2.0 Family Impact Module (PedsQL™) The 36-item PedsQL consists of 6 scales measuring parent self-reported functioning: 1) Physical Functioning (6 items), 2) Emotional Functioning (5 items), 3) Social Functioning (4 items), 4) Cognitive Functioning (5 items), 5) Communication (3 items), 6) Worry (5 items), and 2 scales measuring parent-reported family functioning; 7) Daily Activities (3 items) and 8) Family Relationships (5 items). A 5-point response scale is utilized (0 = never a problem; 4 = always a problem). Items are reverse-scored and linearly transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0) and higher scores indicate better functioning (less negative impact).
Infant blood metabolome | 3 months, 6 months, 9 months, and 1 year
  Newborn blood metabolome as assessed by targeted and untargeted metabolomics from dried blood spots
Alarm Distress Baby scale | 3-4 weeks of age, 2-3 months and 8-10 months of age
  Infant socioemotional development (stress and failure to thrive) will be measured by the Alarm Distress Baby scale. The scale focuses on eight distinctive areas of infant behaviour: facial expression, eye contact, general level of activity, self-stimulation gestures, vocalisations, briskness of response to stimulation, ability to initiate and maintain a relationship and ability to generate and sustain attention. It is used for infants aged 0-24 months and each item is rated from 0 to 4 with the overall score reflecting an interpretation of the baby's behaviour in a given situation. A score of 5 or above is indicative of relational withdrawal.
  A low score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Munk Petersen, MD, PhD, DMSc, Principal Investigator — Center for Klinisk Mikrobiom Forskning, Gastroenheden og Klinisk Mikrobiologisk Afdeling, Hvidovre Hospital
Locations (2):
- Denmark (2):
  - Hvidovre Hospital, Hvidovre, Region Sjælland
  - Center for Klinisk Mikrobiom Forskning, Gastroenheden og Klinisk Mikrobiologisk Afdeling, Hvidovre

IPD SHARING:
Plan to Share IPD: No